CLINICAL TRIAL: NCT01679314
Title: A Prospective, Single Site, Randomized, Controlled, Parallel Group Study in Subjects With Chronic Obstructive Pulmonary Disease (COPD) Stage III and IV Using AlphaCore or Sham (Control, Not Active) as a Prophylactic Treatment
Brief Title: Study to Compare (COPD) Assessment Test in COPD Stage III and IV in a Prophylactic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-001
Record Dates: First submitted 2012-08-15; First posted 2012-09-06 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; non invasive; gammacore
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active AlphaCore device (Active Comparator): AlphaCore active stimulation treatment
  Interventions: Device: AlphaCore device
- Sham AlphaCore device (Sham Comparator): AlphaCore sham device
  Interventions: Device: AlphaCore device

INTERVENTIONS:
Device: AlphaCore device — Each study group will go under the same treatment regimen and assessments.

SUMMARY:
The study will assess the treatment of patients with Chronic Obstructive Pulmonary Disease (COPD) stage III and IV who will self administer the AlphaCore stimulation three times a day over a course of 2 months. Patients will either receive an active AlphaCore device or a Sham device during these two months while not knowing which device they have been provided. At the end of the two months, all patients will be asked to continue in the study for another 2 months to self administer with the active AlphaCore device. Subjects will complete diaries at home on their breathing and quality of life and will return to the clinic monthly for assessment by the investigator.

DETAILED DESCRIPTION:
PERFORMANCE AND SAFETY VARIABLES:

The primary efficacy endpoint for this study is the total Chronic obstructive pulmonary disease (COPD) Assessment Test (CAT) score change from baseline to the 8 week follow-up period comparing the two device groups.

Secondary efficacy endpoints will be the mean difference from baseline to the 8 week follow-up for the following assessments: Medical Research Council (MRC) dyspnoea scale, 6 minutes walking test and Forced Expiratory Volume in one second (FEV1)

Safety Variables:

Each subject will be assessed throughout the study for Adverse Events and at the last visit (4 months) subjects will undergo another physical examination including vital signs and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Diagnosed Chronic obstructive pulmonary disease(COPD) stage III and IV according to Global Initiative for chronic obstructive lung disease (GOLD) guideline
* Forced expiratory volume in one second (FEV 1) < 50%
* Forced expiratory volume in one second (FEV1/Forced expiratory vital capacity (FVC) < 70%
* Signed informed consent form

Exclusion Criteria:

* Participation in other clinical trials (drug or medical device) 30 days prior to start of this study
* Subject is unable to comply with the procedures if the protocol for the study or any other reason judged by the Investigator that could interfere with the study assessment or follow-up
* Has an abscess or other infection or lesion (including lymphadenopathy) at the AlphaCore® treatment site.
* Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Has a history of carotid endarterectomy or vascular neck surgery on the right side.
* Right side or bilateral vagotomy
* Has a recent or repeated history of syncope.
* Has a recent or repeated history of seizures.
* Pregnant or breast feeding women

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias John, MD, Principal Investigator — Praxis für Pneumologie am Asklepios Klinikum Uckermark
Locations (1):
- Praxis fur Pneumologie am Asklepios Klinikum Uckermark, Schwedt, Oder, Germany

IPD SHARING:
Plan to Share IPD: No
No description

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Started | 26 | 28
Completed | 24 | 28
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.2) | 58.0 (7.6) | 59.5 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 17 | 16 | 33
Region of Enrollment [Number; unit: participants]
  Germany | 26 | 28 | 54

OUTCOME MEASURES:

1. Primary Outcome: Chronic Obstructive Pulmonary Disease Assessment Test (CAT) Scores (Quality of Life and Symptoms) Changes Within a Treatment Period and Comparison Between the Two Groups
Description: Chronic obstructive pulmonary disease Assessment Test (CAT) scores (Quality of life and symptoms) changes within a treatment period and comparison between the two groups. Eight (8) questions. The scale is rated from 0 to 5, min = 0, max = 5. Low rates = better, high rates = worse. Mean change in the period 8 weeks versus baseline.
Time Frame: 8 weeks
Population: One patient in the Active AlphaCore device Group missing data at 8 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
units on a scale | -1.3 [-3.2 to 0.6] | -0.9 [-2.7 to 0.8]

2. Secondary Outcome: Change in Borg Dyspnoea Scores
Description: Borg dyspnoea scale (Physical activity test): 0 - 11 (Not at all effected - Extremely effected) The result show the change between the the treatment groups from baseline to week 8
Time Frame: Baseline vs 8 weeks
Population: One subject in the Active AlphaCore device Group missing data at 8 weeks.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Active AlphaCore Device: Active AlphaCore Device Each study group will go under the same treatment regimen and assessments.
- Sham AlphaCore Device: Sham AlphaCore Device Each study group will go under the same treatment regimen and assessments.
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
Scores on a scale | 0.7 (2.0) | 0.4 (1.6)

3. Secondary Outcome: Change 6 Minutes Walking Test
Description: Six minutes walking test: Measure distance (meter) after 6 minutes walk. Change from Baseline between treatment groups
Time Frame: Baseline vs 8 weeks
Population: One patient in the Active AlphaCore group is missing data at week 8
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
Meter | 8.1 (61.5) | 12.6 (55.2)

4. Secondary Outcome: Change in Forced Expiratory Volume (FEV1)
Description: Forced Expiratory Volume (FEV1): Maximum volume that can be exhaled in the first second - after maximum inhalation.
  Change from baseline to week 8 between treatment groups
Time Frame: Baseline vs 8 weeks
Population: One subject in the Active AlphaCore group missing data at week 8
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
Percentage of predicted value
  Baseline | 30.7 (8.8) | 29.7 (8.0)
  Week 8 | 31.0 (9.5) | 31.0 (9.1)

5. Secondary Outcome: Change in EuroQol, 5 Questions and 3 Levels (EQ5D-3L)
Description: The EQ-5D-3L (EuroQoL 5 questions and 3 answering levels) during the run-in period will be compared with the EQ-5D-3L during the treatment period. And treatment period will be compared to open label.
  Rating of questions Level 1 no problems Level 2 some problems Level 3 Significant problems Worst case is 15 points and best case is 5 points using index
Time Frame: Baseline vs 8 weeks
Population: One patient in the Active AlphaCore group is missing data at 8 weeks.
Measure: Number; unit: participants
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
participants
  Mobility-no problem baseline | 7 | 6
  Mobility-no problem week 8 | 8 | 7
  Self Care-no problem baseline | 17 | 21
  Self Care-no problem week 8 | 17 | 22
  Daily Activiies-no problem baseline | 6 | 9
  Daily Activies- no problem week 8 | 4 | 7
  Pain-no problem baseline | 12 | 19
  Pain-no problem week 8 | 15 | 22
  Anxiety-no problem baseline | 12 | 13
  Anxiety-no problem week 8 | 14 | 17

6. Secondary Outcome: Number of Subjects With Adverse Events (AE)
Description: All AEs including but not limited to events reported by the subject or reported in response to an open question by the Clinical Investigator or member of this team, which fall into any of the above definitions must be recorded as an AE in the Case Report Form (CRF) and should include the following information.
  * Brief description of the event (diagnosis)
  * Start date (and time, if relevant)
  * Stop date (and time, if relevant) (or resolution)
  * Severity
  * Action taken regarding the medical device
  * Opinion on causality
  * Seriousness
  * Outcome
Time Frame: Throughout the course of the study (baseline to the 4 month follow-up visit)
Population: All subjects reporting any Adverse Event
Measure: Number; unit: participants
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 26 | 28
participants | 10 | 6

7. Secondary Outcome: Change in Change in EuroQol, 5 Questions and 3 Levels (EQ-5D-3L), Visual Analogue Scale (VAS)
Description: Visual analogue scale (VAS) 0-100 where 0 is the worst imaginable health state and 100 the best imaginable health state
Time Frame: Baseline vs 8 weeks
Population: One patient in the Active AlphaCore group missing data at 8 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Number analyzed (Participants) | 25 | 28
units on a scale
  Baseline | 53.3 (20.0) | 51.6 (16.9)
  8 weeks | 52.8 (18.3) | 55.7 (20.0)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: The first 8 weeks randomized controlled, the last 8 weeks open label
Arm/Group | Active AlphaCore Device | Sham AlphaCore Device
Serious Adverse Events (participants affected / at risk) | 3/26 | 1/28
Other Adverse Events (participants affected / at risk) | 4/26 | 3/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active AlphaCore Device (N=26) | Sham AlphaCore Device (N=28)
Acute COPD exacebartion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalized/Not related
Cartoid stenosis left (Vascular disorders) | 1 (1) | 0 (0) — Hospitalized/Not related
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Hospitalized/Not related
Bronchopneumonia both sides (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalized/Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active AlphaCore Device (N=26) | Sham AlphaCore Device (N=28)
Common cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Infection of the respiratory tract (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No